CLINICAL TRIAL: NCT01232582
Title: Safety and Efficacy of ExAblate MR Guided Focused Ultrasound for the Treatment of Low Back Pain Related to Facet Joint Osteoarthritis
Brief Title: Safety and Efficacy of MRgFUS for the Treatment of Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Nadir Alikacem, Insightec
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FJ001
Record Dates: First submitted 2010-10-28; First posted 2010-11-02 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Lower Back Pain, Facets Joints Osteoarthritis
Keywords: Lower back pain, Facets joints Osteoarthritis
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Exablate treatment — MR guided Focused Ultrasound treatment

SUMMARY:
Chronic pain affects an estimated 50 to 65 million individuals in the US, and its incidence and prevalence is steadily on the rise in correspondence with the increasing longevity of the population. Spinal pain, encompassing lower back, thoracic and neck pain, is a very common type of chronic pain that can greatly reduce quality of life. Facet joint pain is most often associated with facet arthropathy or degenerative arthritis of the joint. This condition develops due to progressive wear and tear caused by the small but repetitive strain of the joints throughout a lifetime. Strain and inflammation can induce fluid distention of the joints which in turn can result in compression of the nerve roots of the joint - the origin of the chronic pain.

Current treatments for facet arthropathy and pain include oral medications, intra-articular injections of anesthetic or steroid medications, energy ablation (e.g. radiofrequency ablation) for denervation, and in some severe cases facet rhizotomy (surgical severing of the nerves).

The ExAblate magnetic resonance guided focused ultrasound system enables noninvasive focal ablation of tissue. Results from feasibility studies, including those from the FDA approved feasibility study (IDE # G050177) have shown the palliative effect of the ExAblate for patients with bone metastases. It is reasonable to assume that this palliative effect of MRgFUS could also translate to the alleviation of facet pain if focused ultrasound beams are directed to the facet joints. The highly-target focal ablation could also diminish the risk of complications that are often associated with other less selective denervation techniques.

The objective of this trial is to evaluate the safety and effectiveness of the ExAblate system and the treatment of pain resulting from facet joint osteoarthritis.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single-arm, phase I study to evaluate the safety and effectiveness of using ExAblate MRgFUS in the treatment of pain resulting from facet joint osteoarthritis.

Patients with chronic LBP associated with one or more lumbar zygapophysial joints that meet all eligibility requirements and have given their written informed consent will be enrolled to the study.

All patients will be treated and followed for 12-months post treatment. A total of 50 patients will be enrolled at up to two clinical sites.

The primary objective of this study is to evaluate incidence and severity of adverse events associated with the ExAblate MRgFUS system used for the treatment of pain resulting from facet joint osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18 and older
2. Patients who are able and willing to give consent and able to attend all study visits
3. Patients who are able to communicate with the treating physician
4. Patients must have chronic LBP attributed to facet joints.
5. Patients with NRS (0-10 scale) LBP average score ≥ 4
6. Patients with chronic LBP for at least 12 months.
7. Patients with Oswestry Disability Questionnaire (ODQ) for LBP score > 40%
8. Targeted Facet joint to be treated is below L2 level

Exclusion Criteria:

1. Patients on dialysis
2. Patients with evidence of lumbosacral radiculopathy on MRI or physical exam findings, including radicular leg pain
3. Patients with RF treatment for LBP within the last 6 months
4. Patients with previous low back surgery
5. Patients who are pregnant
6. Patients with existing malignancy
7. Patients with allergies to relevant anesthetics
8. Patients with motor deficit or any other indication for surgical intervention
9. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations (weight >113 kg)
10. Patients with an acute medical condition (e.g., pneumonia, sepsis) that is expected to hinder them from completing this study.
11. Patients under blood thinners other than Aspirin.
12. Patients with compromised immune system.
13. Patients with unstable cardiac status including:

    * Unstable angina pectoris on medication
    * Patients with documented myocardial infarction less than 40 days prior to protocol enrolment
    * Patients with Severe Congestive Heart Failure, NYHA class 4.
    * Patients on anti-arrhythmic drugs or with uncontrolled and/or untreated arrhythmia status
14. Patients with severe cerebrovascular disease (CVA within last 6 months)
15. Patients with severe hypertension (diastolic BP > 100 on medication)
16. Patients with known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist) including advanced kidney disease
17. Patients with an active infection or severe hematological, neurological, or other uncontrolled disease.
18. Patients unable to communicate with the investigator and staff.
19. Patients who are not able or willing to tolerate the required prolonged stationary position during treatment (approximately 3 hrs.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Adverse events | 12 months
  Evaluate incidence and severity of adverse events associated with the ExAblate MRgFUS system used for the treatment of pain resulting from facet joint osteoarthritis.

SECONDARY OUTCOMES:
Pain Scores on the Numerical Rating Scale | 12 months
  Efficacy will be determined by the level of pain relief (as measured by the Numerical Rating Scale, NRS)
Quality of Life | 12 Months
  Quality of life will be measured by the Oswestry Disability Questionnaire (ODQ), SF-12 Health Survey and pain interference with function (as measured by the Brief Pain Inventory - Interference scale, BPI-QoL)

CONTACTS AND LOCATIONS:
Overall Officials: Sagi Harnof, MD, Principal Investigator — Sheba MC
Locations (2):
- Sheba MC, Ramat Gan, Israel
- St. Mary's Hospital, London, United Kingdom

REFERENCES:
- See also: Sponsor's website — http://www.insightec.com